CLINICAL TRIAL: NCT00208754
Title: Heart Failure in Adult Patients With a History of Congenital Heart Disease.
Status: Terminated | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Wendy M. Book, Principal Investigator, Emory University
Other Study IDs: 0489-2004
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Congenital Heart Defects
Keywords: heart defects; cardiology; adults who have congenital heart defects
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
In today's world of advanced surgery, children born with congenital heart disease (CHD) are surviving into adulthood. However, the surgical procedures these children undergo do not cure the underlying problem and this these children develop other heart problems later in life. Heart failure is the one of the most common heart problems effecting these patients. This heart failure can be seen in both lower pumping chambers of the heart, however, sometimes only one side of the heart is affected. Since there are several congenital heart defects that are now seen in the adult population, an understanding of what causes heart failure in this patient population can help physicians develop better treatments for this condition. The goal of this study is to review the medical records of 350 adult patients with congenital heart disease that has developed heart failure. During this review, we plan to collect information regarding the various treatments utilized in these patients and to determine if there are any common elements regarding the development of heart failure in adult patients with CHD.

DETAILED DESCRIPTION:
In today's world of advanced surgery, children born with congenital heart disease (CHD) are surviving into adulthood. However, the surgical procedures these children undergo do not cure the underlying problem and this these children develop other heart problems later in life. Heart failure is the one of the most common heart problems effecting these patients. This heart failure can be seen in both lower pumping chambers of the heart, however, sometimes only one side of the heart is affected. Since there are several congenital heart defects that are now seen in the adult population, an understanding of what causes heart failure in this patient population can help physicians develop better treatments for this condition. The goal of this study is to review the medical records of 350 adult patients with congenital heart disease that has developed heart failure. During this review, we plan to collect information regarding the various treatments utilized in these patients and to determine if there are any common elements regarding the development of heart failure in adult patients with CHD.

ELIGIBILITY:
Inclusion Criteria:

* Adults who have a history of congenital heart defects

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350
Dates: Start 2004-05; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Book, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Background] Bolger AP, Coats AJ, Gatzoulis MA. Congenital heart disease: the original heart failure syndrome. Eur Heart J. 2003 May;24(10):970-6. doi: 10.1016/s0195-668x(03)00005-8. PMID 12714029
- [Background] Jessup M, Brozena S. Heart failure. N Engl J Med. 2003 May 15;348(20):2007-18. doi: 10.1056/NEJMra021498. No abstract available. PMID 12748317
- [Background] Packer M, Carver JR, Rodeheffer RJ, Ivanhoe RJ, DiBianco R, Zeldis SM, Hendrix GH, Bommer WJ, Elkayam U, Kukin ML, et al. Effect of oral milrinone on mortality in severe chronic heart failure. The PROMISE Study Research Group. N Engl J Med. 1991 Nov 21;325(21):1468-75. doi: 10.1056/NEJM199111213252103. PMID 1944425
- [Background] Deshpande RB, Deodhar LP. Ocular and orbital tumours and tumour-like lesions: a clinico-pathological study of 64 cases. J Postgrad Med. 1977 Apr;23(2):84-8. No abstract available. PMID 614419